CLINICAL TRIAL: NCT03765203
Title: Prospective, Randomized Controlled Trial Using CPV Vignettes to Assess the Clinical Utility of Natera Dd-cfDNA Test to Detect Allograft in Post-Transplant Patients
Brief Title: Utility of a Novel Dd-cfDNA Test to Detect Injury in Renal Post-Transplant Patients
Acronym: QIDNEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Principal Investigator, David Paculdo, John W Peabody, MD PhD, Qure Healthcare, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00030299
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Transplant;Failure,Kidney

STUDY DESIGN:
Intervention Model Description: The study is a pre-post, two round controlled trial of care practices in a nationally representative sample of practicing nephrologists randomly assigned to a control or an intervention arm. All providers will be asked to propose care for a total of 6 CPV simulated patients who are adults aged 30-75; three or more months post-transplant; and presenting with signs, symptoms and laboratory findings suggestive of allograft rejection. Each assessment round will consist of 3 simulated patients. In between assessment rounds, physicians randomized into the intervention arm will receive educational materials on the new allograft rejection test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control participants will care for the same set of CPV patients as the intervention arm, but will not have knowledge of or access to Natera's dd-cfDNA test results. Investigators will compare control participants' clinical recommendations to those in the intervention arm.
  Interventions: Other: Clinical Performance and Value Vignettes
- Intervention (Experimental): Intervention participants will care for the same set of CPV patients as the control arm, but will be educated on and given access to Natera's dd-cfDNA test results. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Diagnostic Test: Natera KidneyScan; Other: Clinical Performance and Value Vignettes

INTERVENTIONS:
Diagnostic Test: Natera KidneyScan — Online educational materials on Natera Kidneyscan (dd-cfDNA) and sample test results for simulated patients
  Arms: Intervention
Other: Clinical Performance and Value Vignettes — Online renal allograft simulated patients
  Other Names: CPVs

SUMMARY:
Detecting allograft injury and rejection is critical to preventing graft loss. The current standard of care (SoC) relies on serum creatinine (SC) and biopsy to monitor for and identify kidney injury earlier. SC has poor specificity and sensitivity and response to rejection is often delayed. Protocol biopsy is more accurate but involves the risk of complications. A more definitive, less invasive method for monitoring injury and early rejection is needed.

We report on the clinical utility of donor-derived cell-free DNA (dd-cfDNA) in transplant recipients' blood, measured using a novel SNP-based mmPCR NGS methodology, to diagnose allograft injury/rejection. In this study, investigators will measure how use of dd-cfDNA changes clinical practice.

DETAILED DESCRIPTION:
Five-year kidney allograft survival rates are estimated to be as low as 71.6%. A leading cause for the high prevalence of graft loss is the delay in detecting allograft injury from active rejection, when early diagnosis and intervention presents the greatest chance of preserving kidney function. Despite the frequent testing called for by care protocols, low levels of injury can go undetected due to the low specificity and sensitivity of current, standard testing methods: checking creatinine and immunosuppressive drug levels. More definitive graft biopsies are an option, but they are invasive, expensive and can even put the patient at risk for graft loss and other complications, making it undesirable as a frequent monitoring test.

Donor-derived cell-free DNA (dd-cfDNA) detected in the blood of transplant recipients has been shown to be a non-invasive diagnostic marker for allograft injury/rejection. Natera, Inc. has recently developed a novel single nucleotide polymorphism (SNP)-based mmPCR NGS methodology to measure dd-cfDNA in kidney transplant recipients for the detection of allograft injury and rejection. As a growing leader in the diagnostic space, Natera has commissioned a randomized controlled trial to determine the clinical utility of its dd-cfDNA detection methodology for practicing nephrologists treating kidney allograft patients. This study is expected to fill a gap in the evidence base on the clinical utility of dd-cfDNA testing for allograft rejection.

The study is a pre-post, two round controlled trial of care practices in a nationally representative sample of practicing nephrologists randomly assigned to a control or an intervention arm. All participants will be asked to propose care for a total of 6 CPV simulated patients who are adults aged 30-75; three or more months post-transplant; and presenting with signs, symptoms and laboratory findings suggestive of allograft rejection. Each assessment round will consist of 3 simulated patients. In between assessment rounds, participants randomized into the intervention arm will receive educational materials on the new allograft rejection test.

Investigators will assess whether practicing nephrologists more effectively identify and manage patients with possible kidney allograft rejection when given access to Natera's novel SNP-based mmPCR-NGS test that measures dd-cfDNA, and, whether those behavioral changes improves patient management and optimizes resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 2 years post-residency but no more than 40 years in practice
* Board-certified in internal medicine
* Completion of a nephrology fellowship
* In a private solo or multi-group practice
* Minimum threshold of 5 post-kidney transplant (KT) patients currently seen monthly
* Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

* Not board certified in internal medicine
* Have practiced as a board-certified physician for less than 2 or greater than 40 years
* See <5 post-transplant patients monthly
* Non-English speaking
* Unable to access the internet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Diagnosis-Treatment | 3 months
  Difference-in-differences regression analysis between the control and the intervention group's identification and treatment of hyperglycemia, as measured by the participants diagnostic and treatment CPV case domain scores. In each domain of a CPV (history, physical exam, workup, diagnosis and treatment), participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum to a high potential score of up to 100% in each domain.

SECONDARY OUTCOMES:
Quality of Care: CPV scores | 3 months
  Difference-in-differences regression analysis between the control and the intervention group's overall quality of care scores. In each CPV case, participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum to a high potential score of up to 100% in each case.
Workup Costs | 3 months
  Difference-in-differences regression analysis between between the control and the intervention group in the average cost of diagnostic tests ordered.

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD PhD, Principal Investigator — President
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No